CLINICAL TRIAL: NCT01805817
Title: Comparison of Levonorgestrel Intrauterine System, Copper T Intrauterine Device and Oral Contraceptives on Life Quality
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cihangir Uzunçakmak, Medical Doctor, OB/GYN, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cuzuncakmak1907
Record Dates: First submitted 2013-02-15; First posted 2013-03-06 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Contraceptive Methods Comparison
Keywords: lipid profile; bleeding scores; menstrual pattern; beneficial; side effects; changes in a year period
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination; drospirenone; Ethinyl Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Levonorgestrel releasing intrauterine device, contraception (Experimental): LNG-IUS - Mirena ®,20μgr, once intrauterine insertion per 5 year, 1 year
  Interventions: Drug: YASMIN® (Drospirenone/Ethinyl Estradiol); Device: The Copper-T is an intrauterine device (IUD); Device: levonorgestrel-releasing system
- YASMIN® (Drospirenone/Ethinyl Estradiol), contraception (Experimental): oral, once a day, 1 year
  Interventions: Drug: YASMIN® (Drospirenone/Ethinyl Estradiol); Device: The Copper-T is an intrauterine device (IUD); Device: levonorgestrel-releasing system
- Copper T 380 A , contraception (Experimental): intrauterine device, once per 10 year, 1 year period
  Interventions: Drug: YASMIN® (Drospirenone/Ethinyl Estradiol); Device: The Copper-T is an intrauterine device (IUD); Device: levonorgestrel-releasing system

INTERVENTIONS:
Drug: YASMIN® (Drospirenone/Ethinyl Estradiol) — oral contraceptive pills
Device: The Copper-T is an intrauterine device (IUD) — intrauterine device for contraception
Device: levonorgestrel-releasing system — intrauterine device
  Other Names: Miirena

SUMMARY:
Oral combined contraceptives(OC) have both progesterone and estrogen inside. Levonorgestrel-releasing intrauterine device(LNG_IUS) has only progestagen.

Copper IUD does not have any hormonal molecule inside.

* Hypothesis is OC has more systemic beneficial or side effects than LNG_IUS or copper IUD. LNG_IUS has more local effects than copper IUD.
* Study reflects the beneficial or side effects of estrogen+progestagen pills and only progestogen inside device.

ELIGIBILITY:
Inclusion Criteria:

* women who desire contraception

Exclusion Criteria:

* Women with large fibroids,abnormal uterine bleeding including heavy menstrual bleeding or using any contraceptive pills during the previous 3 months were excluded from the study. Other exclusion criteria were pelvic inflammatory disease, pregnancy, genital tumor or thromboembolic disease.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Lipid profile (HDL,VLDL,IDL,LDL,Lp(a),VLDL)Lng-ius users, Copper-iud users and combined oral contraceptive users (composite measurement) | Change from Baseline HDL,Very-low-density lipoprotein (VLDL),IDL,Low-density lipoprotein (LDL),Lp(a),VLDL concentrations at 3 months; Baseline to 6 months, Baseline to 12 months of outcome will have assessed
  60 lng-ius users, 60 Copper iud users and 60 combined oral contraceptive users will compared with total lipoprotein, high-density lipoprotein (HDL), low-density lipoprotein (LDL), very-low-density lipoprotein (VLDL), lipoprotein(a) (Lp(a)), intermediate-density lipoprotein (IDL ), HDL subclasses , LDL subclasses , VLDL subclasses ,values at 3-6-12 months follow up.

SECONDARY OUTCOMES:
coagulation parameters(composite measurement) | Change from Baseline aPTT, prothrombin time, INR, D-dimer,factor VIII, fibrinogen, platelet counts values at 3 months; Baseline to 6 months, Baseline to 12 months of outcome will have assessed
  60 lng-ius users, 60 Copper iud users and 60 combined oral contraceptive users will compared with activated partial thromboplastin time (aPTT), prothrombin time, international normalized ratio(INR), D-dimer,factor VIII, fibrinogen, platelet counts values with each other at 3-6-12 months follow up.

OTHER OUTCOMES:
menstrual pattern and bleeding scores(composite measurement) | Change from Baseline pictorial blood scoring system scores at 3 months, Baseline to 6 months, Baseline to 12 months will be assessed
  60 lng-ius users, 60 Copper iud users and 60 combined oral contraceptive users menstrual pattern will be recorded and menstrual bleeding scores will be measured by pictorial blood scoring system and it will be compared with each other at 3-6-12 months follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Haliloglu B, Celik A, Ilter E, Bozkurt S, Ozekici U. Comparison of uterine artery blood flow with levonorgestrel intrauterine system and copper intrauterine device. Contraception. 2011 Jun;83(6):578-81. doi: 10.1016/j.contraception.2010.09.001. Epub 2010 Oct 18. PMID 21570557
- [Background] Sayed GH, Zakherah MS, El-Nashar SA, Shaaban MM. A randomized clinical trial of a levonorgestrel-releasing intrauterine system and a low-dose combined oral contraceptive for fibroid-related menorrhagia. Int J Gynaecol Obstet. 2011 Feb;112(2):126-30. doi: 10.1016/j.ijgo.2010.08.009. Epub 2010 Nov 19. PMID 21092958
- [Background] Mansour D, Gemzell-Danielsson K, Inki P, Jensen JT. Fertility after discontinuation of contraception: a comprehensive review of the literature. Contraception. 2011 Nov;84(5):465-77. doi: 10.1016/j.contraception.2011.04.002. Epub 2011 Jun 8. PMID 22018120
- See also: database for medical publication — http://www.ncbi.nlm.nih.gov/pubmed/?term=lng+ius+combined+oral+contraceptives